CLINICAL TRIAL: NCT03469258
Title: A Phase II Study of Pancreatic Enzyme Replacement (Zenpep) on Completion Rates of Adjuvant Chemotherapy Among Subjects With Resected Pancreatic Ductal Adenocarcinoma
Brief Title: Study of Pancreatic Enzyme Replacement on Completion of Adjuvant Chemotherapy for Resected Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsorship for trial was halted after company acquisition
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, A James Moser, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-450
Record Dates: First submitted 2018-02-15; First posted 2018-03-19 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zenpep (Experimental): * Pancrelipase (Zenpep) will be administered with every meal (breakfast, lunch, dinner) and snack(s), continuously.
  * Participants will begin pancrelipase on the day of enrollment and continue therapy until 1 year after surgery per calendar date
  Interventions: Drug: Pancrelipase

INTERVENTIONS:
Drug: Pancrelipase — Zenpep is a combination of three enzymes (proteins). These enzymes are normally produced by the pancreas and are important in the digestion of fats, proteins, and sugars. Zenpep is used to replace these enzymes when the body does not have enough of its own as a result of surgery and/or pancreatic cancer.
  Other Names: Zenpep

SUMMARY:
This research study is evaluating a study drug to treat pancreatic exocrine insufficiency (PEI) during the first year after the diagnosis of pancreatic cancer while the participant is recovering from surgery and receiving adjuvant treatment.

The study drug involved in this study is:

-Zenpep

DETAILED DESCRIPTION:
The FDA (the U.S. Food and Drug Administration) has approved Zenpep as a treatment option for PEI. Zenpep is a combination of three enzymes (proteins). These enzymes are normally produced by the pancreas and are important in the digestion of fats, proteins, and sugars. Zenpep is used to replace these enzymes when the body does not have enough of its own as a result of surgery and/or pancreatic cancer.

In this research study, the investigators are studying whether Zenpep will improve the ability of patients to complete adjuvant treatment for their pancreatic cancer after surgery to remove their tumor. The investigators are also studying if Zenpep will have an effect on nutrition status and quality of life for pancreatic cancer patients after they have had surgery to remove their tumor.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed pancreatic ductal adenocarcinoma. Variants or mixed histology will be included if the predominant histology is adenocarcinoma.
* Participants must have potentially resectable pancreatic cancer defined as: (1) no detectable metastases (2) signed consent for attempted resection of pancreatic cancer per treating surgeon.
* ECOG performance status ≤2.
* Age >18 years. Participants <18 years old are excluded from this study because subsequent adjuvant therapy is based on therapy guidelines in the adult population.
* Willingness to consider adjuvant therapy following surgical resection of disease, signed in the consent form attestation.
* Ability to understand and willingness to provide written informed consent.
* Pre-operative laboratory values adequate to undergo resection of pancreatic cancer, as defined below:

  * Hemoglobin > 7.0 g/dL;
  * Platelets ≥ 40,000/mL;
  * Creatinine < 2.5 mg/dL or; Creatinine clearance ≥ 20 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.

Exclusion Criteria:

* Pancreatic resection not performed. Intraoperative findings and unforeseen medical exigent circumstances may preclude pancreatic resection. Such outcomes include undetected metastases or vascular involvement, which preclude resection with intent to cure, as well as perioperative medical events including cardiopulmonary complications.
* Final pathology other than pancreatic ductal adenocarcinoma or primary component other than adenocarcinoma.
* Any prior chemotherapy and/or radiation for pancreatic cancer at the time of study enrollment, including neoadjuvant chemotherapy and/or radiation therapy.
* Second malignancy with active disease.
* History of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition to pancrelipase
* Pregnant women are excluded from this study because subsequent adjuvant therapy needed for the primary endpoint is teratogenic. Pancrelipase is category C. Animal reproduction studies have not been conducted on pancrelipase and minimal data is available.
* Participants unable to self-administer pancrelipase.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants who are receiving any other investigational agents.
* Participant unable to tolerate oral nutrition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur James Moser, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Zenpep: * Pancrelipase (Zenpep) will be administered with every meal (breakfast, lunch, dinner) and snack(s), continuously.
  * Participants will begin pancrelipase on the day of enrollment and continue therapy until 1 year after surgery per calendar date
  Pancrelipase: Zenpep is a combination of three enzymes (proteins). These enzymes are normally produced by the pancreas and are important in the digestion of fats, proteins, and sugars. Zenpep is used to replace these enzymes when the body does not have enough of its own as a result of surgery and/or pancreatic cancer.
Period: Overall Study
Arm/Group | Zenpep
Started | 4
Completed | 0
Not Completed | 4
Not completed — Upon surgery, did not meet criteria | 4

BASELINE CHARACTERISTICS:
Population: Patients did not meet pathologic criteria upon surgery. Trial was subsequently terminated by sponsor due to company acquisition.
Arm/Group | Zenpep
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]
Participant must be a candidate for standard of care adjuvant treatment according to their treating

OUTCOME MEASURES:

1. Primary Outcome: Effect of Pancreatic Enzyme Replacement Therapy on the Completion Rate of Adjuvant Chemotherapy and Radiation After Surgery for Early Stage Pancreatic Cancer
Description: Completion, or not, of all doses of chemotherapy and fractions of radiation prescribed by the treating oncologist prior to the start of adjuvant treatment
Time Frame: 40 weeks
Population: Patients did not meet pathologic criteria upon surgery. Trial was subsequently terminated by sponsor due to sponsor acquisition.
Arm/Group | Zenpep
Number analyzed (Participants) | 0

2. Secondary Outcome: Initiation Rate of Adjuvant Treatment for Resected Pancreatic Cancer
Description: Percentage of subjects with resected pancreatic cancer starting adjuvant treatment by postoperative day 84
Time Frame: 84 days after surgery
Population: as for outcome 1
Arm/Group | Zenpep
Number analyzed (Participants) | 0

3. Secondary Outcome: Subject Adherence to Pancreatic Enzyme Replacement Therapy as Determined by Pill Count
Description: Pill count performed by study staff to be compared to subject meal and pill diary to determine percent adherence to prescribed regimen
Time Frame: 52 weeks
Population: as for outcome 1
Arm/Group | Zenpep
Number analyzed (Participants) | 0

4. Secondary Outcome: Subject Adherence to Pancreatic Enzyme Replacement Therapy During Surgery and Adjuvant Treatment for Early Stage Pancreatic Cancer
Description: Pill count performed by study staff will be compared to subject meal and pill diary to determine percent adherence to prescribed regimen
Time Frame: 52 weeks
Population: as for outcome 1
Arm/Group | Zenpep
Number analyzed (Participants) | 0

5. Secondary Outcome: Measure Serum Albumin Levels Before and After Surgery and Adjuvant Treatment for Early Stage Pancreatic Cancer
Description: Quantify serum albumin (g/dl ) to correlate pancreatic enzyme replacement therapy with nutrition status before and after surgery and adjuvant therapy for early stage pancreatic cancer
Time Frame: 52 weeks
Population: as for outcome 1
Arm/Group | Zenpep
Number analyzed (Participants) | 0

6. Secondary Outcome: Measure Body Weight Before and After Surgery and Adjuvant Treatment for Early Stage Pancreatic Cancer
Description: Measure body weight (in kg) at regular intervals throughout study participation to investigate whether pancreatic enzyme replacement therapy improves nutrition status during surgery and adjuvant treatment for early stage pancreatic cancer
Time Frame: 52 weeks
Population: as for outcome 1
Arm/Group | Zenpep
Number analyzed (Participants) | 0

7. Secondary Outcome: Evaluate Quality of Life Before and After Surgery and Adjuvant Treatment for Early Stage Pancreatic Cancer Using the EuroQoL 5 Dimensions 5 Levels (EQ-5D-5L) Questionnaire
Description: Subjects to complete EQ-5D-5L at regular intervals throughout study participation. The scale consists of 5 questions, one each to assess mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each question has answers ranging from No Problems (level 1) to Extreme Problems (level 5). Subjects also to rate their overall health on a given day using the EuroQoL Visual Analog Scale (EQ-VAS) as a part of the EQ-5D-5L, which consists of marking on a visual scale from 0-100 (with 100 being best imaginable health and 0 being worst health imaginable).
Time Frame: 52 weeks
Population: as for outcome 1
Arm/Group | Zenpep
Number analyzed (Participants) | 0

8. Secondary Outcome: Monitor the Incidence and Severity of Complications After Surgery for Early Stage Pancreatic Cancer
Description: Incidence and severity of postoperative complications graded by Clavien-Dindo classification
Time Frame: 84 days after surgery
Population: as for outcome 1
Arm/Group | Zenpep
Number analyzed (Participants) | 0

9. Secondary Outcome: Measure Grip Strength Before and After Surgery and Adjuvant Treatment for Early-stage Pancreatic Cancer
Description: Standard grip strength dynamometer measurements at regular intervals throughout the study
Time Frame: 52 weeks
Population: as for outcome 1
Arm/Group | Zenpep
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 52 weeks after drug initiation and until patient began adjuvant chemotherapy or adjuvant radiation.
Description: The definition of adverse events and/or serious adverse events does not differ from clinicaltrials.gov.
Arm/Group | Zenpep
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Early termination per sponsor leading to small numbers of subjects enrolled. Those subjects who were enrolled did not meet pathologic criteria to remain on study and would have been replaced had the study continued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT03469258/Prot_SAP_000.pdf